CLINICAL TRIAL: NCT06919471
Title: Assessing User Satisfaction and Adherence to an Abbreviated Dietary Tracking App (MySnackTracker) Versus Full-intake Dietary Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0163; NCI-2025-02486 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Dietary Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 2: Fitbit (Experimental): Participants in Group 2, will use the Fitbit food logging app to track their dietary intake. Participants will be asked to log all food and drink intake.
  Interventions: Other: Fitbit
- Group 1: MySnackTracker (Experimental): Participants in Group 1 will use MySnackTracker to track their dietary intake. Participants will be asked to log only high-calorie, low-nutrient food and drinks, or snacks" (for example, cookies, chips and dip, and alcohol). A full list of these foods and drinks is provided in the app.
  Interventions: Other: MySnackTracker App

INTERVENTIONS:
Other: Fitbit — Wear it on wrist
  Arms: Group 2: Fitbit
Other: MySnackTracker App — App to track your dietary intake
  Arms: Group 1: MySnackTracker

SUMMARY:
To learn if a method of abbreviated food tracking (called MySnackTracker) is a reasonable alternative to traditional full-intake food tracking and to compare the adherence to and acceptability of each method.

DETAILED DESCRIPTION:
Primary Objectives The goal of the study is to compare the adherence and acceptability of tracking only high-energy low-nutrient value foods to standard full intake monitoring of diet. We predict that use of the high-energy, low-nutrient-density food tracking app will result in greater adherence to self-monitoring and greater satisfaction with monitoring in comparison to the full intake tracking.

Secondary Objectives Assess the efficacy of the snack tracking app versus standard self-monitoring as measured by changes in the following measures between baseline and follow up; percentage weight change, weight loss self-efficacy scores, food logging self-efficacy scores, GODIN leisure time activity questionnaire scores, Vioscreen tool responses for stages of change for fats and fruit/vegetable intake, daily fruit consumption, daily vegetable consumption, servings of sweets per day, Healthy Eating Index (HEI) Score for calories from solid fats, alcohols, added sugars, HEI empty calories, total drinks of alcohol per day, calories from alcoholic beverages per day, added sugars by available carbohydrates, added sugars by total grams of sugar, calorie intake, carbohydrate intake, fat intake, saturated fatty acid intake, and total sugar intake.

ELIGIBILITY:
Eligibility Criteria

In order to be eligible to participate in this study, an participants must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Access to internet connection, email address, and smartphone able to download the intervention app
* Current or previous participation in one of the following DFI cohorts: PA17-0584 (MERIT Study), Project CHURCH, High Risk Breast Cohort, Mexican-American Cohort, and rural cancer survivors from the Mind Your BEAT study
* Demonstrated ability to read and understand English. The study app is currently only available in English.

Exclusion Criteria

An participant who meets any of the following criteria will be excluded from participation in this study:

* Prisoners
* Anyone currently under 18 years of age
* Cognitively impaired participants
* Pregnant women (assessed by self-report)
* BMI less than 28 or greater than 40
* Self-reported previous or planned bariatric surgery
* Self-reported current or planned use of a GLP-1 agonist medication
* Self-reported current or planned participation in another weight loss intervention
* Cancer participants receiving active treatment
* Anyone currently unable to participate in the research for the duration of the study
* No current motivation to lose weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Basen-Engquist, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org